CLINICAL TRIAL: NCT05043259
Title: Immunogenicity and Safety of the Heterologous Prime-boost Immunization with an Aerosolised Adenovirus Type-5 Vector-based COVID-19 Vaccine (Ad5-nCoV) After Two-dose Priming with an Inactivated SARS-CoV-2 Vaccine in Adults At 18 Years of Age or Above: a Randomised, Open-label, Parallel-controlled Clinical Trial
Brief Title: Heterologous Prime-boost Immunization with an Aerosolised Adenovirus Type-5 Vector-based COVID-19 Vaccine (Ad5-nCoV) After Priming with an Inactivated SARS-CoV-2 Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT127
Record Dates: First submitted 2021-09-13; First posted 2021-09-14 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Aerosolised COVID-19 vaccine; Recombinant Ad5 Vector; Inactivated Vaccine; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Inactivated vaccine group (Active Comparator): Subjects who have been vaccinated with two doses of inactivated SARS-CoV-2 vaccine will receive one dose of inactivated SARS-CoV-2 vaccine
  Interventions: Biological: inactive SARS-CoV-2 vaccine (Vero cell)
- Low dose aerosolized Ad5-nCoV group (Experimental): Subjects who have been vaccinated with two doses of inactivated SARS-CoV-2 vaccine will receive one dose of the low dose of aerosolized Ad5-nCoV.
  Interventions: Biological: Low dose aerosolized Ad5-nCoV
- High dose aerosolized Ad5-nCoV group (Experimental): Subjects who have been vaccinated with two doses of inactivated SARS-CoV-2 vaccine will receive one dose of the high dose of aerosolized Ad5-nCoV.
  Interventions: Biological: High dose aerosolized Ad5-nCoV

INTERVENTIONS:
Biological: inactive SARS-CoV-2 vaccine (Vero cell) — This vaccine contains 600 SU of SARS-CoV-2 antigen, which is produced by Sinovac Research & Development Co., Ltd. 0.5 ml / bottle.
  Arms: Inactivated vaccine group
Biological: Low dose aerosolized Ad5-nCoV — This vaccine is produced by CanSino Biologics Inc. It is a liquid dosage form, 0.1 ml / dose, contains 1×10^10 virus particles of recombinant replication defective human type 5 adenovirus expressing SARS-CoV-2 S protein, aerosol inhalation.
  Arms: Low dose aerosolized Ad5-nCoV group
Biological: High dose aerosolized Ad5-nCoV — This vaccine is produced by CanSino Biologics Inc. It is a liquid dosage form, 0.2 ml / dose, contains 2×10^10 virus particles of recombinant replication defective human type 5 adenovirus expressing SARS-CoV-2 S protein, aerosol inhalation.
  Arms: High dose aerosolized Ad5-nCoV group

SUMMARY:
This is a randomized, open-label, parallel-controlled study to evaluate the safety and immunogenicity of heterologous prime-boost immunization with an aerosolised adenovirus type-5 vector-based COVID-19 vaccine (Ad5-nCoV) after priming with an inactivated SARS-CoV-2 vaccine in adults at 18 years of age or above. 420 healthy subjects aged over or equal to 18 years whom have received two doses of inactivated SARS-CoV-2 vaccines within the last 3~9 months, will be recruited in this study. Eligible participants will be randomized at a 1:1:1 ratio to receive a booster dose of inactive SARS-CoV-2 vaccine or a low dose of aerosolized Ad5-nCoV or a high dose of aerosolized Ad5-nCoV. The occurrence of adverse events within 28 days and serious adverse events within 6 months after vaccination will be observed. In addition, blood samples will be collected on the day 0 before and day 7, 14, 28 and month 3, 6, and 12 after the booster vaccination. Each subject will remain in this study for approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Health subjects aged ≥18 years, completed two dose of inactive SARS-CoV-2 vaccine in the past 3-9 months.
* The subject can provide with informed consent and sign informed consent form (ICF).
* The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the 12-month follow-up of the study.
* No nasal or oral diseases, such as acute rhinitis (sinusitis), allergic rhinitis, oral ulcer, sore throat, etc.
* Axillary temperature ≤ 37.0℃
* Individuals who are in good health condition at the time of entry into the trial as determined by medical history, physical examination and clinical judgment of the investigator and meet the requirements of immunization

Exclusion Criteria:

* have the medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
* be allergic to any component of the research vaccines, or used to have a history of hypersensitivity or serious reactions to vaccination.
* suffering from abnormal pulmonary function such as asthma, chronic obstructive pulmonary disease and pulmonary fibrosis.
* suffering from more serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension and uncontrollable medication.
* have symptoms of upper respiratory tract infection.
* women with positive urine pregnancy test, pregnant or breast-feeding, or have a pregnancy plan within six months.
* have acute febrile diseases and infectious diseases.
* have severe chronic diseases or condition in progress cannot be smoothly controlled, such as asthma, diabetes, thyroid disease
* congenital or acquired angioedema / neuroedema.
* have the history of urticaria 1 year before receiving the investigational vaccine.
* have asplenia or functional asplenia.
* have thrombocytopenia or other coagulation disorders (which may cause contraindications for intramuscular injection).
* have needle sickness.
* have the history of immunosuppressive therapy, anti-allergy therapy, cytotoxic therapy or inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, and acute corticosteroid therapy without dermatitis) over the past 6 months.
* have received blood products within 4 months before injection of investigational vaccines.
* have received another investigational product within one month before injection of investigational vaccine.
* have received attenuated vaccine within 1 month before injection of investigational vaccine.
* under anti-tuberculosis treatment.
* not be able to follow the protocol, or not be able to understand the informed consent according to the researcher's judgment, due to various medical, psychological, social or other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions within 14 days after the booster dose. | Within 14 days the booster dose
  Incidence of adverse reactions within 14 days after vaccination.
GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 14 after the booster dose. | On day 14 after the booster dose
  GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 14 after the vaccination.

SECONDARY OUTCOMES:
Incidence of adverse events within 0-28 days after the booster dose. | within 28 days after the booster dose.
  Incidence of adverse events (AE) within 0-28 days after the booster vaccination.
Incidence of serious adverse events (SAE) till the 12 months after the booster dose. | within 12 months after the booster dose.
  Incidence of serious adverse events (SAE) till the 12 months after booster vaccination.
GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 7 and 28 after the booster dose. | on day 7 and 28 after the boost vaccination.
  GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 7 and 28 after the booster dose.
Fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus on day 14 after the booster vaccination. | on day 14 after the last dose of vaccination.
  Fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus, as compared to baseline, on day 14 after the booster vaccination.
GMT, fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus at month 3, 6, and 12 after the booster dose. | at month 3, 6, and 12 after the boost vaccination.
  GMT, fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus at month 3, 6, and 12 after the booster dose.
GMT, fold increase and seroconversion of binding antibodies against SARS-CoV-2 RBD on day 7, day 14, day 28 after the booster dose. | on day 7, day 14, day 28 after the booster vaccination.
  GMT, fold increase and seroconversion of binding antibodies against SARS-CoV-2 S and N protein measured by ELISA on day 7, day 14, day 28 after the booster vaccination.
GMT, fold increase and seroconversion of binding antibodies against SARS-CoV-2 RBD at month 3, 6, and 12 after the booster dose. | at month 3, 6, and 12 after the booster vaccination.
  GMT, fold increase and seroconversion of binding antibodies against SARS-CoV-2 S and N protein measured by ELISA at month 3, 6, and 12 after the booster vaccination.
The levels of IFN- γ、IL-2 and IL-13 secreted by specific T cells on day 7 and 14 after the booster vaccination. | on day 7 and 14 after the booster vaccination.
  The levels of IFN- γ、IL-2 and IL-13 secreted by specific T cells on day 7 and 14 after the booster vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Xin Li, PhD, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Donghai County Center for Diseases Control and Prevention, Lianyungang, Jiangsu, China

REFERENCES:
- [Derived] Jin L, Tang R, Wu S, Guo X, Huang H, Hou L, Chen X, Zhu T, Gou J, Zhong J, Pan H, Cui L, Chen Y, Xia X, Feng J, Wang X, Zhao Q, Xu X, Li Z, Zhang X, Chen W, Li J, Zhu F. Antibody persistence and safety after heterologous boosting with orally aerosolised Ad5-nCoV in individuals primed with two-dose CoronaVac previously: 12-month analyses of a randomized controlled trial. Emerg Microbes Infect. 2023 Dec;12(1):2155251. doi: 10.1080/22221751.2022.2155251. PMID 36503413
- [Derived] Li JX, Wu SP, Guo XL, Tang R, Huang BY, Chen XQ, Chen Y, Hou LH, Liu JX, Zhong J, Pan HX, Shi FJ, Xu XY, Li ZP, Zhang XY, Cui LB, Tan WJ, Chen W, Zhu FC; CanSino COVID-19 Study Group. Safety and immunogenicity of heterologous boost immunisation with an orally administered aerosolised Ad5-nCoV after two-dose priming with an inactivated SARS-CoV-2 vaccine in Chinese adults: a randomised, open-label, single-centre trial. Lancet Respir Med. 2022 Aug;10(8):739-748. doi: 10.1016/S2213-2600(22)00087-X. Epub 2022 May 20. PMID 35605625